CLINICAL TRIAL: NCT05558540
Title: Spinal Cord Stimulation for Intractable Chronic Lower Abdominal Neuropathic Pain Caused by Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Velja Mijatovic (Other)
Collaborators: Boston Scientific Group (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Velja Mijatovic, Professor Doctor, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL76287.018.21
Record Dates: First submitted 2022-09-15; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: All women participating in the trial will receive a SCS. Women will first undergo a trial period of 14 days. If succesful (>50% pain reduction), women will receive a permanently implanted SCS. The follow-up period will enclose 12 months. There is an aimed sample size of 15 participants. However, due to financial limitations, inclusion will stop after 10 women have been succesfully implanted with a permanent SCS.
Masking Description: Due to the nature of the intervention, masking is not possible. All participants will receive a SCS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Implantation with spinal cord stimulator (Experimental): Women participating in the trial will receive a spinal cord stimulator (SCS). Women will first undergo a trial implantation period of 14 days. When the trial period is considered successfull (at least 50 percent reported pain reduction) women will receive definitive placement of the SCS. Normal lead placement( bilateral TH8-12) and different stimulation types will be used (FAST, subthresholdand/orCombination). When participating in the trial, women will be asked to complete a set of questionnaires on several occasions, i.e. at baseline, 3 months after implantation, 6 months after implantation and 12 months after implantation.
  Interventions: Device: spinal cord stimulator

INTERVENTIONS:
Device: spinal cord stimulator — By continuous electrical stimulation of the nerve causing endometriosis-related pain, painful inputs to the spinal cord and brain can be reduced or even eliminated. The electrical stimulation is performed by the spinal cord stimulator (SCS).
  Other Names: neuromodulation

SUMMARY:
Endometriosis is a chronic, inflammatory disease where endometrium-like tissue is present outside the uterus. Nerve cells in the proximity of this tissue express cytokine receptors causing a signaling cascade. This results in active cross-talk between endometriosis and nerves, causing pelvic pain. Other symptoms associated with endometriosis are cyclical such as dysmenorrhea and dysuria, and non-cyclical such as dyspareunia. Despite adequate disease management, women can still experience endometriosis-related pain. A recent development proven to be efficient in treatment of neuropathic pain, is Spinal Cord Stimulation (SCS). It is also thought to be effective in the treatment of visceral pain. Several studies found Spinal Cord Stimulation (SCS) to be effective in the reduction of endometriosis-related pelvic pain. However, scientific evidence on the efficacy of SCS in visceral pain is limited.

DETAILED DESCRIPTION:
Endometriosis is an estrogen-dependent gynaecologicalcondition characterized by the presence and growth of ectopic endometrial tissue. This tissue stimulates the infiltration of immune cells such as macrophages andmast cells into the peritoneal cavity. Both the immune cells and the endometriotic tissue secrete cytokines which create an inflammatory microenvironment. Nerve cells located in the proximity of endometriosis lesions express cytokine receptors which stimulate a cascade of signalling kinases within the nerve. This results in an active cross-talk between endometriosis and nerves causing endometriosis associated pain.

Because of the chronic nature of endometriosis, treatment can be challenging difficult. It consists of three pillars: hormonal therapy, surgery and conventional pain management. Despite adequate disease management, women with endometriosis can still experience endometriosis-associated chronic pelvic pain. This might suggest that the pathology was either an incidental finding, or that other mechanisms continue to generate pain without the need for a peripheral input. One study proposed that central sensitization may be involved mechanistically in the development and maintenance of endometriosis-related pain. The hypothesis was that persistent nociceptive input from endometriotic tissues might result in increased responsiveness among dorsal horn neurons processing input from the affected viscera and pelvic tissues [1].

When standard endometriosis treatment is insufficient in the suppression of endometriosis-related pelvic pain, spinal cord stimulation (SCS), an accepted treatment option for neuropathic pain, could be a potential treatment.This hypothesis was substantiated by several (case) studies. However, they stated that studies on SCS for treatment of visceral pain is limited and made a call for action to broaden this knowledge

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal woman aged ≥ 18 years
* Patients with endometriosis/ adenomyosis confirmed at surgery macroscopically and without options for further surgical treatment.
* Patients with at least one of the endometriosis related pain symptoms: dysmenorrhea, pelvic pain or dyspareunia. With a mean pain NRS of at least 5 (scale 0-10).
* The pain complaints are therapy resistant (including hormonal, medical and/or surgical options).
* Refractory pain; before neuromodulation patient has tried: Paracetamol, NSAIDs, Anti neuropathic pain therapy, TENS.
* The patient meets all the inclusion criteria for the implantation of a neurostimulation system as typically utilized in the study center.
* Neurologic exam without marked motor deficit.
* Subject has been screened by a multi-disciplinary panel including a psychologist and deemed suitable for implantation
* Subject is able and willing to comply with the follow-up schedule and protocol
* Subject is able to provide written informed consent

Exclusion Criteria:

* Female subject of childbearing potential is pregnant/nursing or plans to become pregnant during the course of the study.
* The presence of malignancy
* Subject currently has an active implantable device including ICD, pacemaker, spinal cord stimulator or intrathecal drug pump
* Subject is unable to operate the device
* Previous Neurostimulation therapy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with female reproductive organs can be diagnosed with endometriosis. Endometriosis does not occur in the male population. Therefore, only women can be included in the trial. Patients identifying as female but without female reproductive organs can unfortunately not participate in the trial.
Enrollment: 15 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain severity at 6 month follow-up | 6 months
  An aimed pain reduction of at least 30% or 2 points reduction in mean NRS pain score (0-10). This is measured using a pain diary.

SECONDARY OUTCOMES:
Change in Mean pain from baseline until 12 month follow-up | 12 months
  Measured using a pain diary, women report their pain score expressed with the Numeric rating scale (NRS) pain scores) 3 times a day for 3 days at baseline, 3-and 12-months post implant.
Patient's global impression of change | 12 months
  Measured using the PGIC questionnaire. Dichotomous (better or improved versus not better or improved) at baseline,3-6-and 12-months post implant.
Change in quality of life | 12 months
  Measured using the EHP-30 questionnaire at baseline, 3-6-and 12-months post implant. Each scale was transformed on a range from 0 to 100. A score of "0" stands for best possible health status. A score of "100" stands for worst possible health status.
Change in quality of life | 12 months
  Measured using the SF-36 questionnaire at baseline, 3-6-and 12-months post implant. Scores are divided between 8 domains and calculated. They range from 0 to 100, and are compiled as a percentage. The higher the score, the more favorable the health state.
Change in fatigue | 12 months
  Measured using the shortened fatigue questionnaire (SFQ) at baseline, 3-6-and 12-months post implant. Scores can range between 4 and 28. The higher the score, the more severe the fatique.
Change in Pain Catastrophizing Scale | 12 months
  Measured using the PCS questionnaire. Measured at baseline, 3-6-and 12-months post implant. A score between 0 and 52 can be calculated. The higher the score, the more severe the patient catastrophizes her pain.
Change in Central Sensitization Inventory | 12 months
  Measured using the CSI questionnaire. Measured at baseline, 3-6-and 12-months post implant. A score between 0 and 100 can be calculated. A score between 0-29 stands for subclinical central sensitization syndrome (CSS). A score between 30 and 39 for mild SCC. A score between 40 and 49 for moderate SCC. A score between 50 and 59 for severe SCC. A score between 60-100 for extreme SCC.
Change in pain medication use | 12 months
  Assessed using a questionnaire. Women are asked on their possible use of pain medication at baseline, 3-month, 6-month and 12-month follow up. Use of pain medication is compared between the follow-up moments.
Lost working days | 6 months
  Measured using the EHP-30 at baseline and at 6 months post implant. Asked using part A of the modular questionnaire. A score between 0 and 100 can be calculated. The higher the score, the higher the impact of endometriosis on working life.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bajaj P, Bajaj P, Madsen H, Arendt-Nielsen L. Endometriosis is associated with central sensitization: a psychophysical controlled study. J Pain. 2003 Sep;4(7):372-80. doi: 10.1016/s1526-5900(03)00720-x. PMID 14622679
- [Derived] van Haaps AP, Kallewaard JW, Bieze M, Erwteman M, Nap A, Hollmann MW, Schreurs AMF, Mijatovic V. Spinal-Cord Stimulation for Intractable, Visceral Pain Associated With Endometriosis: Positive Results of a Feasibility Study. Neuromodulation. 2025 Dec 3:S1094-7159(25)01143-2. doi: 10.1016/j.neurom.2025.10.067. Online ahead of print. PMID 41335088